CLINICAL TRIAL: NCT00664209
Title: Helicobacter Pylori Eradication and Motor Fluctuations in Parkinson's Disease
Brief Title: Treating H. Pylori in Parkinson's Patients With Motor Fluctuations
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Prevalence of H Pylori in the study population was much lower than anticipated
Sponsor: University of California, Los Angeles (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Jeff Bronstein, Professor of Neurology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJJF Clinical Discovery 2007; 441437-JB-58330
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease; Helicobacter Infections; Motor Fluctuations
Keywords: Parkinson's disease; levodopa; Helicobacter pylori
MeSH Terms: conditions — Parkinson Disease; Helicobacter Infections | interventions — Amoxicillin; Omeprazole; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active-placebo (Other): These subject receive treatment with active triple therapy followed by treatment with placebo therapy.
  Interventions: Drug: clartihromycin, amoxicillin, and omeprazole; Drug: placebo
- Placebo-active (Other): These subject receive treatment with placebo therapy followed by treatment with active triple therapy.
  Interventions: Drug: clartihromycin, amoxicillin, and omeprazole; Drug: placebo

INTERVENTIONS:
Drug: clartihromycin, amoxicillin, and omeprazole — clarithromycin 500mg - i PO BID x10 days; amoxicillin 1gm - i PO BID x10 days; omeprazole 10mg - i PO BID x10 days
  Other Names: Biaxin, Prilosec
Drug: placebo — placebo therapy

SUMMARY:
The purpose of this study is to determine whether treatment of H. pylori (an infection of the stomach) improves treatment effectiveness in patients with Parkinson's disease and motor fluctuations.

DETAILED DESCRIPTION:
Previous investigations have demonstrated that treatment of Helicobacter pylori with antibiotics leads to improved absorption and pharmacokinetics of levodopa. This may potentially benefit patients with Parkinson's disease who have motor fluctuations, specifically excessive "off" time, when their levodopa is not working to control symptoms. We seek to identify the frequency of H. pylori infection in this population using standard lab assays and determine whether eradication with standard triple therapy results in improved clinical response to medication.

ELIGIBILITY:
Inclusion criteria:

* Adults diagnosed with idiopathic Parkinson's disease, Hoehn & Yahr stage 2-4 in the "off" state, with no other concomitant neurologic diseases.
* Stable (≥30 days) Parkinson's disease therapy, with demonstrable medication efficacy, but with wearing off phenomenon present between levodopa doses (average off time ≥3 hours off time/day).
* Levodopa therapy required; Any formulation (e.g. Sinemet, Sinemet CR, Stalevo) is acceptable. Parkinson's disease treatment may also include any of the following medications or classes: non-ergot dopamine agonists, COMT inhibitors, MAO-B inhibitors, amantadine, anticholinergics.
* Positive for H. pylori IgG Ab by serum ELISA (before inclusion in randomized treatment arms).

Exclusion criteria:

* Current abdominal pain, unexplained nausea/vomiting, or gastrointestinal bleeding.
* History of gastric cancer, peptic ulcer, duodenal ulcer, or other gastric or duodenal lesions.
* History of previous gastric surgery.
* History of previous brain surgery for Parkinson's disease.
* Family history of gastric cancer.
* Prior treatment for H. pylori+ status.
* Recent use (previous 4 weeks) of proton-pump inhibitor, amoxicillin, or clarithromycin.
* Allergy or sensitivity to penicillin, amoxicillin, clarithromycin, or omeprazole.
* Use of drugs affecting gastric motility (e.g. domperidone, metoclopramide).
* Inability to tolerate or participate in testing in the morning in an "off" state.
* Inability to communicate effectively with study personnel in English.
* Pregnancy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff M Bronstein, MD, PhD, Principal Investigator — UCLA Neurology
Locations (1):
- UCLA Neurology, Los Angeles, California, United States

REFERENCES:
- [Background] Belhoussine-Idrissi L, Boedeker EC. Helicobacter pylori infection: treatment. Curr Opin Gastroenterol. 2002 Jan;18(1):26-33. doi: 10.1097/00001574-200201000-00005. PMID 17031226
- [Background] Pierantozzi M, Pietroiusti A, Brusa L, Galati S, Stefani A, Lunardi G, Fedele E, Sancesario G, Bernardi G, Bergamaschi A, Magrini A, Stanzione P, Galante A. Helicobacter pylori eradication and l-dopa absorption in patients with PD and motor fluctuations. Neurology. 2006 Jun 27;66(12):1824-9. doi: 10.1212/01.wnl.0000221672.01272.ba. PMID 16801644
- [Background] Pierantozzi M, Pietroiusti A, Galante A, Sancesario G, Lunardi G, Fedele E, Giacomini P, Stanzione P. Helicobacter pylori-induced reduction of acute levodopa absorption in Parkinson's disease patients. Ann Neurol. 2001 Nov;50(5):686-7. doi: 10.1002/ana.1267. No abstract available. PMID 11706979
- [Background] Pierantozzi M, Pietroiusti A, Sancesario G, Lunardi G, Fedele E, Giacomini P, Frasca S, Galante A, Marciani MG, Stanzione P. Reduced L-dopa absorption and increased clinical fluctuations in Helicobacter pylori-infected Parkinson's disease patients. Neurol Sci. 2001 Feb;22(1):89-91. doi: 10.1007/s100720170061. PMID 11487216
- [Background] Wolle K, Malfertheiner P. Treatment of Helicobacter pylori. Best Pract Res Clin Gastroenterol. 2007;21(2):315-24. doi: 10.1016/j.bpg.2006.11.001. PMID 17382279

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 64 enrolled, 13 positive for H. Pylori were screened for motor fluctuations (wearing off of the benefits of levodopa).
Groups:
- Active: Those with significant wearing-off were to be assigned to arms, and received open-label triple eradication therapy (standard of care) per physician decision because the screen yield was too low to test effect size between arms.
  ---- Clarithromycin 500mg - i PO BID x10 days; Amoxicillin 1gm - i PO BID x10 days; Omeprazole 10mg - i PO BID x10 days
Period: Motor Fluctuations Screen
Arm/Group | Active
Started | 13
Completed | 6
Not Completed | 7
Not completed — Negative for motor fluctuation | 7
Period: Study Treatment Period
Arm/Group | Active
Started | 6
Completed | 0
Not Completed | 6
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Active: H. Pylori positive participants screened for eligibility to a treatment assignment.
Arm/Group | Active
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 62.4 [51 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: "Off" Time
Description: Average total daily "off" time (measured by patient symptom diaries) in hours
Time Frame: 2 months
Population: Participants did not return symptom diaries
Groups:
- Active: Standard treatment with active triple therapy
Arm/Group | Active
Number analyzed (Participants) | 0

2. Secondary Outcome: Improvement in UPDRS Total Scores
Description: The Unified Parkinson Disease Rating Scale (UPDRS) is a rating tool to follow the longitudinal course of Parkinson's Disease. It is made up of the 1) Mentation, Behavior, and Mood, 2) ADL and 3) Motor sections. These are evaluated by interview. Some sections require multiple grades assigned to each extremity. A total of 199 points are possible. 199 represents the worst (total) disability), 0--no disability.
Time Frame: 2 months
Population: Subjects H pylori positive with greater than 4 hrs off time/day and completing the UDPRS
Arm/Group | Active
Number analyzed (Participants) | 0

3. Secondary Outcome: Improvement in UDPRS Part III
Description: Improvement in UDPRS Part III (Motor) scores ("on" and "off") UPDRS III is the result of a motor examination with the scores 0-108. A decrease in the scores means improvement
Time Frame: 2 months
Population: Subjects H pylori positive with greater than 4 hrs off time/day and completing the UDPRS
Arm/Group | Active
Number analyzed (Participants) | 0

4. Secondary Outcome: Improvement in Quality of Life as Assessed by PDQ-39
Description: The Parkinson's Disease Questionnaire (PDQ)-39 contains 39 questions addressing how often patients have experienced difficulties due to having PD in the preceding month. Items are scored from 0 (never) to 4 (always). Lower scores indicate better quality of life.
Time Frame: 2 months
Population: Subjects H pylori positive with greater than 4 hrs off time/day and completing the PDQ-29
Arm/Group | Active
Number analyzed (Participants) | 0

5. Secondary Outcome: Participants With Side Effects From Study Treatment
Description: Side effects profile
Time Frame: 2 months
Population: All subjects receiving H. pylori treatment
Measure: Number; unit: participants
Arm/Group | Active
Number analyzed (Participants) | 6
participants | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Screening yield was much lower than anticipated based on the literature which prohibited completion of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No